CLINICAL TRIAL: NCT04152876
Title: Functional Genomics of Rare Genetic Diseases: Realization of Innovative Tools With High Diagnostic Power
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Neuromed IRCCS (Other)
Collaborators: Institute of Genetics and Biophysics CNR (Unknown)
Responsible Party: Principal Investigator, Diego Centonze, Head of Neurology Unit, Neuromed IRCCS
Other Study IDs: PON MISE n. F/050011/01/X32
Record Dates: First submitted 2019-11-04; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Rare Diseases
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples for DNA extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients with rare disease
- controls: Healthy parents and relatives

SUMMARY:
The project aims to improve the understanding of a significant group of rare diseases both from a genetic/diagnostic and clinical/experimental point of view and aims to develop one or more diagnostic protocols.

The study will be conducted through the application of complementary experimental strategies, ranging from the clinical, genetic and molecular characterization of the pathology to the search for rare variants and the development of cellular disease models.

DETAILED DESCRIPTION:
1. Clinical evaluation of patients and relatives
2. High throughput analysis of genetic variants in genome exomes
3. Genotype-phenotype association testing
4. Identification of genetic risk variants for rare diseases

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by: SLA, Incontinentia Pigmenti type II, Rett Syndrome, Paget Disease, Pompe Disease, Immunodeficiency, Centromeric instability and Facial anomalies, Cortical malformations and malignant epileptic encephalopathies

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be selected from the Center for rare diseases of the IRCCS Neuromed, and at IGB CNR according to specific inclusion criteria. Approximatey 300 subjects, recruited with a family-based approach, will be included in the study.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-10-31 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Identification of genetic variants responsible for rare diseases | Two years
  Analysis of exome sequencing data; annotation of genetic variants; selection of variants present in cases and absent in controls

CONTACTS AND LOCATIONS:
Overall Officials: Diego Centonze, MD, Principal Investigator — Head of Neurology Unit
Locations (1):
- IRCCS Neuromed, Pozzilli, Italy